CLINICAL TRIAL: NCT02575170
Title: Intravenous Amino Acid Infusion in Mothers Before and During Cesarean Delivery: Effects on Maternal and Neonatal Temperature
Brief Title: Amino Acid Infusion in Mothers Before and During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Krishna Pokharel, Dr (MD), B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 599/068/069
Record Dates: First submitted 2015-10-04; First posted 2015-10-14 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Hypothermia
Keywords: amino acid; cesarean delivery; hypothermia
MeSH Terms: conditions — Hypothermia | interventions — amino-acid, glucose, and electrolyte solution; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amino acid (Experimental): Intravenous infusion of amino acid solution started approximately one hour prior to spinal anaesthesia after recording the baseline vital parameters. Each patient in experimental group received a total of 200 ml at 2 ml/kg/min.
  Interventions: Drug: Amino acid solution
- Ringer's Lactate solution (Placebo Comparator): Intravenous infusion of Ringer's lactate solution started approximately one hour prior to spinal anaesthesia after recording the baseline vital parameters. Each patient in experimental group received a total of 200 ml at 2 ml/kg/min.
  Interventions: Drug: Ringer's lactate solution

INTERVENTIONS:
Drug: Amino acid solution — a balanced mixture of 18 pure crystalline amino acids, eight of which are essential amino acids
  Other Names: Alamin SN ®, Albert D Limited, Kolkata, India
  Arms: Amino acid
Drug: Ringer's lactate solution — 200 ml of Ringer's lactate solution
  Other Names: RINGER LACTATE SOLUTION ALBERT DAVID
  Arms: Ringer's Lactate solution

SUMMARY:
Introduction: Intravenous infusion of amino acids during cesarean delivery in mothers and neonates improves neonatal growth. Amino acid before and during anesthesia also prevents hypothermia and associated untoward effects.

Method: After ethical approval, this prospective randomized double blind controlled study is being conducted in the university hospital of BPKIHS. Seventy six parturients (ASA 1 & 2) undergoing cesarean delivery without fetal distress, intrauterine growth retardation, congenital malformation or premature labor will be enrolled.

For a period starting from approximately one hour prior to spinal anesthesia, Group 1 and Group 2 patients will receive 200 ml of amino acid and lactated ringers solution respectively at 2 ml/kg/hr. The ambient operating room temperature will be maintained near 23º C. No heating methods will be applied apart from covering with a blanket.

Primary outcome measure will be neonatal rectal temperature at 0, 5 and 10 min after birth. Secondary outcome measures will be APGAR scores and suckling reflex in the newborn, change in rectal temperature relative to baseline and discomfort related to cold sensation in the mother and the occurrence of shivering both in the mother and newborn.

DETAILED DESCRIPTION:
Review of literature:

Hypothermia is common during peri-operative period (1). It can lead to shivering (2), sympathetic stimulation (3), ischemic cardiac events (3), coagulation disturbances (4,5) delayed recovery from anesthesia (6,7), altered immune system with impaired wound healing (8,9) and prolonged hospitalization (9).

Amino acid infusion before and during surgery is known to prevent peri-operative hypothermia as a result of increased thermogenesis (10,11) without additional sympatho-adrenal activity (12). The mechanism is based on nutrient induced thermogenesis; i.e., nutrient intake, especially proteins and amino acids, stimulates resting energy expenditure and heat production (13). This effect is more pronounced during general anesthesia than neuraxial block (14). It has also been proved that amino acid infusion before and/or during anesthesia and surgery decreases intra-operative blood loss (15), improves peri-operative recovery (16) and shortens the duration of hospital stay (17).

The safety of intravenous amino acid infusion during cesarean delivery was long ago established (18,19).While maternal intravenous administration of amino-acids led to increased levels of amino acids in maternal venous blood and fetal umbilical cord blood plasma, there was no increase in fetal uptake of amino acids.

The safety of amino acid in the first day of life after delivery has also already been proved (20,21). It has been used to achieve positive protein balance in the immediate postoperative period in neonates undergoing abdominal surgery (20). Aggressive therapy of intravenous amino acid in preterm infants during 12 hrs to two weeks after birth enhanced their growth and improved their nutritional status during hospitalization (21).

Rationale of the study:

One way to prevent the development of hypothermia during anesthesia is to stimulate endogenous heat production. Energy expenditure increases after ingestion or infusion of nutrients. The amount of energy expended over baseline, or thermic effect of food mainly represents the energy cost of nutrient absorption, handling, and storage. Among the different nutrients, proteins elicit the largest increase in energy expenditure and heat production.

Previous studies have found that intravenous amino acid infusions exert enhanced thermogenic effects during general anesthesia (10) The mechanism behind this phenomenon is not fully understood, although nutrient intake stimulates energy expenditure, and hence heat production, in the awake state (13). The administration of proteins/amino acids in awake individuals results in an approximately 20% increase in whole-body heat content and a significant increase in body temperature (22,23).

Since amino acid transfer across the placenta depends upon its concentration in maternal blood (21,24), the investigators hypothesize that by increasing its concentration in the maternal blood, the amino acid level in newborn will be increased. The amino acid induced increased thermogenesis in the mother is likely to increase maternal temperature and thus fetal temperature. Also amino acids that have crossed the placenta may increase thermogenesis in the fetus, further enhancing neonatal temperature.

Research design and methodology:

After getting approval from the institutional research ethics committee and written informed consent, this prospective randomized double blind study was conducted in the University hospital of B P Koirala Institute of Health Sciences (BPKIHS). Parturients belonging to American Society of Anesthesiologists physical status I and II scheduled for elective cesarean delivery were enrolled. Pregnancy with fetal distress, intrauterine growth retardation, congenital malformation or premature labor were excluded.

With the help of computer generated random numbers, each consecutive eligible patients scheduled for cesarean delivery were assigned to one of the two groups to receive 200 ml of intravenous amino acid (Active drug) (n=38) or nutrient free standard ringers lactate solution (active comparator) (n=38) at 2 ml/kg/hr approximately one hour before spinal anesthesia. Amino acid solution used was a balanced mixture of 18 pure crystalline amino acids, eight of which are essential amino acids (Alamin SN ®, Albert D Limited, Kolkata, India).

On the pre-anesthetic visit one day prior to surgery, all the patients were explained about the nature of the study and the various questions to be asked during the study. Approximately 90 minutes prior to surgery, each patient was taken to the pre-operative room inside the operation theater. Heart rate, respiratory rate, rectal temperature and SpO2 were monitored continuously and non invasive blood pressure every five minutes. To maintain blinding, all the infusion bags were covered with an opaque plastic sheet and labelled as 'infusion bag' and hanged on the infusion stand near the patient by an anesthetist not involved in the management or data collection thereafter. Intravenous infusion of amino acid solution or ringer's solution was started approximately one hour prior to spinal anesthesia after recording the baseline vital parameters. Each patient received a total of 200 ml at 2 ml/kg/min. Both the patients and the assessor were unaware of the group assignment.

After one hour of infusion, each patient was transferred to the operating room. The ambient temperature of the operating room was maintained near 23°C. The monitoring of non invasive blood pressure, heart rate, respiratory rate, oxygen saturation (SpO2) and rectal temperature were continued at the same intervals. Spinal anesthesia was induced with 2 ml of 0.5% bupivacaine at L 3-4 inter-space applying aseptic precautions with the patient in the lateral position. After administration of spinal anesthesia, both groups received Ringers solution 15-20 ml/kg/hr maintained at ambient temperature via a separate venous access. All the patients were covered with a blanket, but no other heating methods were applied. Amino acid infusion were continued till the completion of 200 ml the solution contained in the infusion bag.

The maternal rectal temperature were recorded before infusion (baseline), prior to spinal block, at the time of delivery, at half an one hour after spinal block, and at the end of infusion of 200 ml of study solution. At the end of surgery, each mother was asked about her perception of cold and its related discomfort on a 0-2 subjective scale (0= No perception, 1= Tolerable perception, 2=Intolerable perception).

The rectal temperature and APGAR scores were assessed at 0, 5 and 10 minutes and suckling reflex at 10 minutes of the birth of baby. The occurrence of shivering and duration of hospital stay were noted for both the mother and baby.

Primary outcome parameters was the neonatal rectal temperature at 0, 5 and 10 minutes after birth. Secondary outcome parameters included neonatal APGAR scores at 0, 5 and 10 minutes after birth, the number of newborn having suckling reflex; number of neonates who developed shivering within 10 minutes after birth; change in maternal rectal temperature relative to baseline at various time points during study drug infusion, maternal temperature at the time of delivery during intraoperative period; number of mothers developing cold sensation related discomfort during the intra-operative period; number of mothers who developed shivering during intra-operative period.

Previous report showed that the mean rectal temperature of new born immediately after delivery following spinal anaesthesia was 37.7°C. (22) With the help of STATA, it was estimated that a sample size of 26 in each group could achieve a power of 95% to detect a difference of 0.5 °C (with common standard deviation of 0.5) in the outcome measure of new born rectal temperature, assuming type 1 error of 0.05.

For the secondary outcome, the sample size was calculated using online statistical calculator G power (R) version 3.0.1. Cohen d was used to calculate the effect size based on the findings of a previous study.(14) The mean final core temperature 90 min after induction of spinal anaesthesia was 35.8 (SEM 0.1)°C in the saline group and 36.6 (0.1)°C in the amino acid group.(14) It was estimated that a sample size of 34 in each group could achieve a power of 80% to detect an effect size of 0.69 in the outcome measure of maternal core body temperature, assuming type 1 error of 0.05. We enrolled 38 patients in each group to compensate for dropout cases and shifting from normality in data distribution.

ELIGIBILITY:
Inclusion Criteria:

* Parturients belonging to American Society of Anesthesiologists physical status I and II scheduled for elective cesarean delivery were enrolled.

Exclusion Criteria:

* Pregnancy with fetal distress, intrauterine growth retardation, congenital malformation or premature labor were excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
neonatal rectal temperature | 0 min after delivery
neonatal rectal temperature | 5 min after delivery
neonatal rectal temperature | 10 min after delivery

SECONDARY OUTCOMES:
APGAR score of newborn | 0 min, 5 min, 10 min after birth
number of newborn with adequate suckling reflex | 10 min after birth
  absent or present
scale assessing the discomfort related to cold sensation in mother | intraoperative period during spinal anesthesia
  0= No perception, 1= Tolerable perception, 2=Intolerable perception
number of mothers who developed shivering | intraoperative period during spinal anesthesia
length of hospital stay of mother | up to 72 hours
length of hospital stay of newborn | up to 72 hours
change in maternal rectal temperature compared to baseline | before infusion (baseline) and 1 hour
maternal rectal temperature | at the time of delivery during intraoperative period (usually within 30 minutes)
change in maternal rectal temperature compared to baseline | before infusion (baseline) and at one hour after spinal block
change in maternal rectal temperature compared to baseline | before infusion (baseline) and at the end of infusion of 200 ml of study solution
number of neonates who developed shivering | during the first 10 min after birth

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Pokharel, MD, Study Chair — B.P. Koirala Institute of Health Sciences
Locations (1):
- B P Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

REFERENCES:
- [Background] Sessler DI. Mild perioperative hypothermia. N Engl J Med. 1997 Jun 12;336(24):1730-7. doi: 10.1056/NEJM199706123362407. No abstract available. PMID 9180091
- [Background] Sessler DI, Rubinstein EH, Moayeri A. Physiologic responses to mild perianesthetic hypothermia in humans. Anesthesiology. 1991 Oct;75(4):594-610. doi: 10.1097/00000542-199110000-00009. PMID 1928769
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Valeri CR, Feingold H, Cassidy G, Ragno G, Khuri S, Altschule MD. Hypothermia-induced reversible platelet dysfunction. Ann Surg. 1987 Feb;205(2):175-81. doi: 10.1097/00000658-198702000-00012. PMID 3813688
- [Background] Rohrer MJ, Natale AM. Effect of hypothermia on the coagulation cascade. Crit Care Med. 1992 Oct;20(10):1402-5. doi: 10.1097/00003246-199210000-00007. PMID 1395660
- [Background] Lenhardt R, Marker E, Goll V, Tschernich H, Kurz A, Sessler DI, Narzt E, Lackner F. Mild intraoperative hypothermia prolongs postanesthetic recovery. Anesthesiology. 1997 Dec;87(6):1318-23. doi: 10.1097/00000542-199712000-00009. PMID 9416715
- [Background] Heier T, Caldwell JE, Sessler DI, Miller RD. Mild intraoperative hypothermia increases duration of action and spontaneous recovery of vecuronium blockade during nitrous oxide-isoflurane anesthesia in humans. Anesthesiology. 1991 May;74(5):815-9. doi: 10.1097/00000542-199105000-00003. PMID 1673591
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Sellden E, Brundin T, Wahren J. Augmented thermic effect of amino acids under general anaesthesia: a mechanism useful for prevention of anaesthesia-induced hypothermia. Clin Sci (Lond). 1994 May;86(5):611-8. doi: 10.1042/cs0860611. PMID 8033514
- [Background] Sellden E, Branstrom R, Brundin T. Preoperative infusion of amino acids prevents postoperative hypothermia. Br J Anaesth. 1996 Feb;76(2):227-34. doi: 10.1093/bja/76.2.227. PMID 8777102
- [Background] Sellden E, Lindahl SG. Amino acid-induced thermogenesis reduces hypothermia during anesthesia and shortens hospital stay. Anesth Analg. 1999 Dec;89(6):1551-6. doi: 10.1097/00000539-199912000-00045. PMID 10589647
- [Background] Jequier E. The influence of nutrient administration on energy expenditure in man. Clin Nutr. 1986 Nov;5(4):181-6. doi: 10.1016/0261-5614(86)90022-1. PMID 16831767
- [Background] Kasai T, Nakajima Y, Matsukawa T, Ueno H, Sunaguchi M, Mizobe T. Effect of preoperative amino acid infusion on thermoregulatory response during spinal anaesthesia. Br J Anaesth. 2003 Jan;90(1):58-61. PMID 12488380
- [Background] Widman J, Hammarqvist F, Sellden E. Amino acid infusion induces thermogenesis and reduces blood loss during hip arthroplasty under spinal anesthesia. Anesth Analg. 2002 Dec;95(6):1757-62, table of contents. doi: 10.1097/00000539-200212000-00053. PMID 12456453
- [Background] Saitoh Y, Kaneda K, Tokunaga Y, Murakawa M. Infusion of amino acid enriched solution hastens recovery from neuromuscular block caused by vecuronium. Br J Anaesth. 2001 Jun;86(6):814-21. doi: 10.1093/bja/86.6.814. PMID 11573589 (Retraction: PMID 30579399 Br J Anaesth. 2019 Jan;122(1):155)
- [Background] Xing A, Wan B, Zeng W. [Biochemical effects of maternal intravenous and intra-amniotic infusion of amino-acids on fetal blood]. Hua Xi Yi Ke Da Xue Xue Bao. 1994 Mar;25(1):98-102. Chinese. PMID 8070785
- [Background] Ronzoni S, Marconi AM, Cetin I, Paolini CL, Teng C, Pardi G, Battaglia FC. Umbilical amino acid uptake at increasing maternal amino acid concentrations: effect of a maternal amino acid infusate. Am J Obstet Gynecol. 1999 Aug;181(2):477-83. doi: 10.1016/s0002-9378(99)70581-8. PMID 10454703
- [Background] Reynolds RM, Bass KD, Thureen PJ. Achieving positive protein balance in the immediate postoperative period in neonates undergoing abdominal surgery. J Pediatr. 2008 Jan;152(1):63-7. doi: 10.1016/j.jpeds.2007.05.042. Epub 2007 Sep 17. PMID 18154902
- [Background] Wang C, Han LY, Zhang LJ, Wang DH. [Effect of aggressive nutritional support on preterm infants during hospitalization]. Zhonghua Er Ke Za Zhi. 2011 Oct;49(10):771-5. Chinese. PMID 22321185
- [Background] Brundin T, Wahren J. Influence of protein ingestion on human splanchnic and whole-body oxygen consumption, blood flow, and blood temperature. Metabolism. 1994 May;43(5):626-32. doi: 10.1016/0026-0495(94)90206-2. PMID 8177052
- [Background] Brundin T, Wahren J. Effects of i.v. amino acids on human splanchnic and whole body oxygen consumption, blood flow, and blood temperatures. Am J Physiol. 1994 Mar;266(3 Pt 1):E396-402. doi: 10.1152/ajpendo.1994.266.3.E396. PMID 8166259
- [Background] Regnault TR, de Vrijer B, Battaglia FC. Transport and metabolism of amino acids in placenta. Endocrine. 2002 Oct;19(1):23-41. doi: 10.1385/ENDO:19:1:23. PMID 12583600
- [Background] Fallis WM, Hamelin K, Symonds J, Wang X. Maternal and newborn outcomes related to maternal warming during cesarean delivery. J Obstet Gynecol Neonatal Nurs. 2006 May-Jun;35(3):324-31. doi: 10.1111/j.1552-6909.2006.00052.x. PMID 16700681
- [Derived] Pokharel K, Subedi A, Tripathi M, Biswas BK. Effect of amino acid infusion during cesarean delivery on newborn temperature: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 Mar 31;21(1):267. doi: 10.1186/s12884-021-03734-4. PMID 33789610